CLINICAL TRIAL: NCT02150330
Title: Effects of Dehydroepiandrosterone Supplementation on Cumulus Cells Gene Expression Under Controlled Ovarian Hyper-stimulation in Patients With Diminished Ovarian Reserve
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National YangMing University (Unknown)
Responsible Party: Principal Investigator, vghtpe user, Peng-Hui Wang, M.D. Ph D., Department of Obstetrics and Gynecology, Taipei Veterans General Hospital, Taipei, Taiwan, ROC, Taipei Veterans General Hospital, Taiwan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS13-CT11-17
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Dehydroepiandrosterone; DHEAS; Gene Expression of Cumulus Cells.; Ovarian Hyper-stimulation Protocol.; Artificial Reproduction Technology.
Keywords: Dehydroepiandrosterone; DHEAS; Gene expression of cumulus cells.; Folliculogenesis.; Oocyte maturation.; Ovarian hyper-stimulation protocol.; Artificial reproduction technology.
MeSH Terms: interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DHEAS in DOR Group (Active Comparator): Additional usage of DHEAS supplement in patients with DOR under ovarian hyper-stimulation protocol.
  Interventions: Drug: Dehydroepiandrosterone (DHEAS)
- Normal Control (Active Comparator): Patients under ovarian hyper-stimulation protocol. No DHEAS supplement.
  Interventions: Drug: Dehydroepiandrosterone (DHEAS)
- Shame DOR Group (Active Comparator): Patients with DOR under ovarian hyper-stimulation protocol. No DHEAS supplement.
  Interventions: Drug: Dehydroepiandrosterone (DHEAS)

INTERVENTIONS:
Drug: Dehydroepiandrosterone (DHEAS)
  Other Names: DHEAS

SUMMARY:
Diminished ovarian reserve (DOR) is one the challenge in the field of artificial reproductive technology (ART) while there is still no effective resolution of this disorder. In patents with DOR, the pregnancy rate is about only 2-4%. Eventually, patients with DOR turn to adapt children instead. In recent studies, dehydroepiandrosterone (DHEAS) supplement might play a role in reverse diminished ovarian reserve and improve the prognosis of ART. Cumulus cells, formed cumulus-oocyte complex (COC) with oocyte, play a important role in folliculogenesis, oocyte maturation, oocyte meiosis and ovulation. Growing evidences disclose there are crosstalks between oocyte and cumulus cells as paracrine regulations. Aberration the crosswalks between oocytes and cumulus cells would be associated with poor prognosis of folliculogenesis and further pregnancy outcomes. In patients under ovarian hyper-stimulation protocol, the assessment of cumulus cells might be reliable indicators of folliculogenesis, embryo development, pregnancy rate and pregnancy outcomes. These genes (indicators), such as Hyaluronan synthase（HAS2), Versican (VCAN), Thrombospondin 1 (THBS1), Runt-related transcription factor 2 (RUNX2), Chromobox homolog 3 (CBX3),Tripartite motif-containing 28 (TRIM28), B-cell lymphoma 2 (BCL2)，BCL2-associated X protein (BAX). This study was assess the gene expressions of cumulus cells after the DHEAS supplement in patients with DOR under ovarian hyper stimulation protocol.

DETAILED DESCRIPTION:
This study was designed as a prospective case-control study to assess the gene expression of cumulus cells after DHEAS supplement. Patients with diminished ovarian reserve under ovarian hyper-stimulation protocol were evaluated at Kaoshiung Veteran General Hospital from January 1, 2013 through October 31, 2013. Approval for the study was obtained from the hospital's ethic committee, and informed consent was obtained from all patients (VGHKS13-CT11-17)

ELIGIBILITY:
Inclusion Criteria:

* DOR: antral follicle count (AFC) less than 5, AntiMullerian hormone (AMH) less than 1.0 ng/ml, and previous total retrieved oocyte less than 5.
* Normal Control: antral follicle count (AFC) equal to or more than 5, AntiMullerian hormone (AMH) equal to or more than 1.0 ng/ml, and previous total retrieved oocyte equal to or more than 5.

Patient provided signed informed consent.

Exclusion Criteria:

* Patient who has the allergic history or contraindication to DHEAS usage.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Gene expressions of culumuls cells under ovarian hyper-stimulation protocol. | The 3 or 5 days after oocyte retrieval.
  Assessment of gene expressions of cumulus cells, including Hyaluronan synthase (HAS2), Versican (VCAN), Thrombospondin 1(THBS1), Runt-related transcription factor 2 (RUNX2), Chromobox homolog 3 (CBX3), Tripartite motif-containing 28 (TRIM28), B-cell lymphoma 2 (BCL2), BCL2-associated X protein (BAX).

SECONDARY OUTCOMES:
Pregnancy outcomes were compared with diminished ovarian reserve and normal control groups after DHEAS supplement. | 2 to 4 weeks after embryo transfer.
  The successful pregnancy outcome is defined as intrauterine gestational sac with positive fetal heart activity on the sonogram.

CONTACTS AND LOCATIONS:
Overall Officials: KuanHao Tusi, M.D., Principal Investigator — Kaohsuing Veteran General Hospital; PengHui Wang, M.D.,Ph D, Study Chair — Taipei Veteran General Hospital, National YangMing University
Locations (1):
- Taipei Veteran General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Tsui KH, Lin LT, Chang R, Huang BS, Cheng JT, Wang PH. Effects of dehydroepiandrosterone supplementation on women with poor ovarian response: A preliminary report and review. Taiwan J Obstet Gynecol. 2015 Apr;54(2):131-6. doi: 10.1016/j.tjog.2014.07.007. PMID 25951716
- [Derived] Tsui KH, Lin LT, Horng HC, Chang R, Huang BS, Cheng JT, Wang PH. Gene expression of cumulus cells in women with poor ovarian response after dehydroepiandrosterone supplementation. Taiwan J Obstet Gynecol. 2014 Dec;53(4):559-65. doi: 10.1016/j.tjog.2014.09.003. PMID 25510701